CLINICAL TRIAL: NCT06066112
Title: Study on the Bioequivalence of Amisulpride Orally Disintegrating Tablets (200 mg) in Chinese Healthy Subjects Under Single Dose, Randomized, Open, Two Formulation, Two Sequence, Two Cycle, Double Crossover, Fasting, and Postprandial Conditions
Brief Title: Study on the Bioequivalence of Amisulpride Orally Disintegrating Tablets in Human Body
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HQ-0124-BE01
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Bioequivalence; Schizophrenia
Keywords: amisulpride orally disintegrating tablets
MeSH Terms: conditions — Schizophrenia | interventions — Drug Evaluation; Long-Term Synaptic Depression; Amisulpride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting state (Experimental): The subjects fasted overnight for at least 10 hours, and an indwelling needle was buried before administration. On the morning of administration, one test formulation (T) or one control formulation (R) was administered on an empty stomach, and the start time of administration was recorded. After administration, the oral cavity and medication container should be checked to ensure the correct use of the medication. Do not drink water from 1 hour before medication to 1 hour after medication (except for 20ml of water moistened with the test formulation and 240 mL of water from the control formulation). Control drinking water from 1 hour to 4 hours after medication, and drink freely at other times. Fasting within 4 hours after medication. After medication, keep the upper body upright for 4 hours. The meal time on the day of the two cycles of medication is roughly the same.
  Interventions: Drug: Drug: Test (T) Amisulpride orally disintegrating tablets (200mg). Produced and supplied by Zezheng (Shanghai) Biotechnology Co., Ltd.
- Fed state (Experimental): Before administration, subjects were placed with an indwelling needle and fasted overnight for at least 10 hours before consuming a high-fat meal. They started eating a high-fat meal 30 minutes before taking the medication on the morning of the day of administration. Control drinking water from 1 hour to 4 hours after taking the medication, and drink freely at other times. Fasting within 4 hours after taking the medication. After medication, keep the upper body upright for 4 hours. The meal time on the day of the two cycles of medication is roughly the same.
  Interventions: Drug: Drug: Test (T) Amisulpride orally disintegrating tablets (200mg). Produced and supplied by Zezheng (Shanghai) Biotechnology Co., Ltd.

INTERVENTIONS:
Drug: Drug: Test (T) Amisulpride orally disintegrating tablets (200mg). Produced and supplied by Zezheng (Shanghai) Biotechnology Co., Ltd. — Randomly assign to TR or RT sequence groups based on a predetermined random table and receive the corresponding study drug according to the corresponding administration sequence.
  Other Names: Reference (R) Amisulpride tablets (200mg). Produced and supplied by Zezheng (Shanghai) Biotechnology Co., Ltd.

SUMMARY:
The experiment adopts a single center, randomized, open, single dose, two cycle, and double crossover design. The subjects were randomly divided into TR and RT groups. In the first cycle, they received the test or control formulation on an empty stomach or after a meal. After a cleaning period, they entered the second cycle and received the control or test formulation in the same state. The cleaning period between the two cycles was 7 days.

ELIGIBILITY:
Inclusion Criteria:

* 1. Chinese male or female subjects aged ≥ 18 years old (including 18 years old);

  2. Weight: Male ≥ 50 kg, female ≥ 45 kg, and body mass index (BMI) between 19.0 and 26.0 kg/m2 (including boundary values, BMI=weight (kg)/height 2 (m2));

  3. During the screening period, the vital signs, physical examination, laboratory examination, and electrocardiogram of the subjects were found to be normal or abnormal, and were determined by the researchers to be clinically insignificant;

  4. All fertile subjects agree to take appropriate and effective physical contraception measures for themselves and their partners from the screening period (female subjects from 2 weeks before screening) to the end of the experiment, and to take effective physical contraception and/or medication contraception measures within 6 months after the end of the experiment, without any plans for sperm or egg donation;

  5. The subjects fully understand the purpose, nature, and potential adverse reactions of the experiment, understand and follow the research process, voluntarily participate, and sign an informed consent form;

  6. Those who are able to communicate well with researchers and understand and comply with the requirements of this study.

Exclusion Criteria:

* 1. Those with a past or existing history of the following diseases or chronic/severe illnesses, including but not limited to the cardiovascular system, digestive system, urogenital system, respiratory system, blood system, endocrine system, immune system, mental nervous system, skeletal system, etc., that researchers believe are still clinically significant; Especially for subjects with gastrointestinal dysfunction, peptic ulcer, gastrointestinal surgery, and other diseases that affect drug absorption, distribution, metabolism, and excretion;

  2. Screening subjects who have undergone surgery within the first 3 months, or who plan to undergo surgery during the study period, or who have undergone surgery that affects drug absorption, distribution, metabolism, and excretion;

  3. There is a history of food and drug allergies that researchers have determined to be clinically significant; Or known allergies to sulfamethoxide or its excipients, or a history of other allergic diseases (asthma, urticaria, eczema dermatitis);

  4. Previous or existing history of vascular edema or peripheral edema;

  5. Screening for individuals with blurred vision, visual abnormalities, diplopia, or fundus lesions within the first 14 days; 6. Individuals with oral diseases such as oral ulcers during the screening period;

  7. Previous or existing xerostomia patients;

  8. People with positive results of any test for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or treponema pallidum antibody (TP Ab);

  9. Screening for individuals with a history of drug abuse or positive urine drug abuse screening within the previous 12 months;

  10. Regular drinkers within the first 6 months of screening, i.e. those who consume an average of more than 14 units of alcohol per week (1 unit ≈ 285 mL of beer with an alcohol content of 3.5%, 25 mL of spirits with an alcohol content of 40%, or 85 mL of wine with an alcohol content of 12%), or those who cannot dispose of alcohol 48 hours before administration until the end of the study, or those who have tested positive for alcohol breath during the screening period; 11. Smoking an average of more than 5 cigarettes per day in the first 3 months of screening; Or those who cannot give up smoking 48 hours before administration until the end of the study;

  12. Receive blood transfusion or use blood products within 3 months before screening; Those who have donated blood or experienced significant bleeding (greater than 400 mL, except for blood loss during normal physiological periods in females) within 3 months before the first administration, or plan to donate blood or blood components during the study period or within 1 week after the end of the study;

  13. Screening subjects who have participated or are currently participating in other clinical trials within the first 3 months (drug clinical trials are defined as those who have used clinical research drugs);

  14. Screening subjects who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, health products, and functional vitamins within the previous 14 days; Or those who have received vaccines within 2 weeks before screening or those who have vaccination plans during the trial period;

  15. Those who have special dietary requirements, cannot accept a unified diet, and comply with corresponding regulations; Or those who consume beverages (coffee, tea) or food (animal liver) rich in xanthine during the experiment, or consume fruits or juice such as grapefruit, grapefruit, mango, etc. that may affect drug metabolism;

  16. Individuals with rare genetic diseases such as lactose or galactose intolerance, primary lactase deficiency, or glucose galactose malabsorption; 17. Pregnant or lactating female subjects; Female reproductive age subjects who engage in sexual activity without effective contraceptive measures within 14 days prior to signing the informed consent form;

  18. Those with difficulty swallowing;

  19. Patients with poor vascular puncture conditions, inability to tolerate venous puncture, or those with needle and blood fainting;

  20. Other subjects deemed unsuitable by the researchers to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-10-07 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Cmax | 48 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | 48 hours
  Area under the drug concentration-time curve from time 0 to the last accurately measurable concentration at sample collection time t
Area under the plasma concentration versus time curve (AUC0-∞) | 48 hours
  Area Under the Plasma Drug Concentration-Time Curve from Time 0 to Infinite Time

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University Phase I Clinical Research Center, Qingdao, Shandong, China